CLINICAL TRIAL: NCT07383025
Title: Mavacamten Post-marketing Surveillance in Patients With Obstructive Hypertrophic Cardiomyopathy (oHCM) in Japan
Brief Title: Mavacamten Post-marketing Surveillance in Patients With Obstructive Hypertrophic Cardiomyopathy in Japan
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV027-1081
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy (oHCM)
Keywords: Obstructive hypertrophic cardiomyopathy (oHCM)
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with obstructive hypertrophic cardiomyopathy receiving mavacamten treatment
  Interventions: Drug: Mavacamten

INTERVENTIONS:
Drug: Mavacamten — According to the product label

SUMMARY:
The purpose of this study is to assess the real-world effectiveness and safety of mavacamten in patients with obstructive hypertrophic cardiomyopathy (HCM) receiving mavacamten in Japan

ELIGIBILITY:
Inclusion Criteria:

• All obstructive hypertrophic cardiomyopathy (oHCM) patients who initiate treatment with Mavacamten of the approved indications at medical institutions in Japan during enrollment period will be enrolled in this regulatory post-marketing surveillance (PMS) study

Exclusion Criteria:

• Participants receiving Mavacamten for an off-label indication will be excluded from this PMS study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults diagnosed with obstructive hypertrophic cardiomyopathy (oHCM) who initiate mavacamten treatment at medical institutions in Japan
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and/or serious AEs (SAEs) | Up to 52 weeks
Actions taken after adverse events (AEs) and/or serious AEs (SAEs) | Up to 52 weeks
Outcome of adverse events (AEs) and/or serious AEs (SAEs) | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- CMIC Co., Ltd, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts